CLINICAL TRIAL: NCT02388867
Title: Predictive Role of Matrix Metalloproteinases for the Outcome of Surgical Revascularization in Patients With Critical Limb Ischemia
Brief Title: Matrix Metalloproteinases in Patients With Critical Limb Ischemia Undergoing Surgical Revascularization
Acronym: ROMAMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Prof. Raffaele Serra, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ER.ALL.2014.10.A
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Critical Limb Ischemia; Extracellular Matrix Alteration; Peripheral Revascularisation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Polytetrafluoroethylene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Intervention: Polytetrafluoroethylene (PTFE) bypass grafting.
  Interventions: Procedure: Polytetrafluoroethylene (PTFE) bypass grafting.
- Group II (Experimental): Intervention: Autogenous vein bypass grafting.
  Interventions: Procedure: Autogenous vein bypass grafting

INTERVENTIONS:
Procedure: Polytetrafluoroethylene (PTFE) bypass grafting. — Polytetrafluoroethylene (PTFE) bypass grafting. Patients will undergo bypass procedure using PTFE graft : the inflow vessel may be the femoral artery or the iliac artery; the outflow vessel may be the popliteal artery or the anterior tibial artery.
  Arms: Group I
Procedure: Autogenous vein bypass grafting — Autogenous vein bypass grafting. Patients will undergo Bypass procedure using autogenous veins (the great saphenous vein or the small saphenous vein or a composite bypass using great and small saphenous vein ). The inflow vessel may be represented by the femoral artery or the popliteal artery; the outflow vessel may be the anterior tibial artery or the posterior tibial artery or the peroneal artery.
  Arms: Group II

SUMMARY:
In the present study the investigators will evaluate MMPs. serum levels variations in patients affected by critical limb ischemia, before and after lower limb surgical revascularization through venous or prosthetic bypass.

DETAILED DESCRIPTION:
Recent clinical studies showed an association between Peripheral Artery Disease (PAD) and circulating levels of Matrix Metalloproteinases (MMPs), especially MMP-2, MMP-9, MMP-8 and MMP-10, compared with healthy controls. A recent study showed the association between MMP-10 serum levels and severity and poor outcome in patients affected by Critical Limb Ischemia (CLI).

Also, MMPs seems to be involved in intimal hyperplasia and constrictive remodeling, both responsible of restenosis after surgical treatment of atherosclerotic lesions.

Intimal hyperplasia is a thickening of the tunica intima resulting in narrowing of the vessel lumen.

Elevated tissue levels of MMP-2 and MMP-9 have been identified in pig models of vein bypass grafts, temporally coinciding with the period of Smooth Muscle Cells (SMC) migration and neointimal formation.

In the present study the investigators want to evaluate MMP-1; MMP-2, MMP-9, MMP-8 and MMP-10 serum levels variations in patients affected CLI, before and after lower limb surgical revascularization through venous or prosthetic bypass in order to assess their role in predicting the surgical outcome of these procedures.

Patients with CLI will be randomized to receive lower limb surgical revascularization through autogenous venous (Group I) or prosthetic bypass (using synthetic polytetrafluoroethylene - PTFE- ) (Group II).

Patients enrolled in the present study will be followed through clinical and ultrasonographic examination at 1, 3, 6, 12 and 24 months. At the same time points MMPs plasma levels (by means of blood sampling through venipuncture) will be evaluated. Clinical, Instrumental and Laboratory data then will be matched.

ELIGIBILITY:
Inclusion Criteria:

* patients with CLI stage III-IV according to the Fontaine's classification

Exclusion Criteria:

* Patients with evidence of systemic sepsis, known neoplastic disease or any established generalized inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
MMPs evaluation | 24 months
  MMPs plasma levels will be evaluated during follow up.